CLINICAL TRIAL: NCT04730427
Title: A Phase 1b Study to Investigate the Safety and Preliminary Efficacy of GX-I7 in Patients With COVID-19
Brief Title: Safety and Preliminary Efficacy Study of GX-I7 in Patients With COVID-19
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Genexine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GX-I7-COV-009
Record Dates: First submitted 2021-01-20; First posted 2021-01-29 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — efineptakin alfa

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GX-I7 (Experimental): GX-I7
  Interventions: Drug: GX-I7
- GX-I7 vehicle (Placebo Comparator): GX-I7 vehicle
  Interventions: Drug: GX-I7 vehicle

INTERVENTIONS:
Drug: GX-I7 — Recombinant human interleukin-7 hybrid Fc
  Other Names: Efineptakin alfa; rhIL-7-hyFc; NT-I7; TJ107
  Arms: GX-I7
Drug: GX-I7 vehicle — Formulation buffer of recombinant human interleukin-7 hybrid Fc
  Arms: GX-I7 vehicle

SUMMARY:
This study is a phase 1b clinical trial to investigate the safety and preliminary effects of a single dose of a test drug or placebo to the subjects who has diagnosed as COVID-19 infection.

DETAILED DESCRIPTION:
This study is a phase 1b clinical trial to investigate the safety and preliminary effects of a single dose of a test drug or placebo to the subjects who has diagnosed as COVID-19 infection.

Study design: prospective, randomized, placebo-controlled, single-blind, single-center

ELIGIBILITY:
Key Inclusion Criteria:

1. Subjects who have been confirmed to be COVID-19 corresponding to mild cases of severity categorization classified by FDA through polymerase chain reaction (PCR) test or virus gene test (sequencing) and who can be available to be administered within seven days from the date of manifestation.
2. Subjects who are or will be inpatient.

Key Exclusion Criteria:

1. Patients with symptoms of moderate or higher in the severity classification presented by FDA have evidence of lower respiratory tract infection in their imaging findings or need supplemental oxygen therapy or mechanical respiration (ie, non-invasive ventilation, invasive mechanical ventilation, extracorporeal membrane oxygenation, etc)
2. Subjects with infectious diseases such as bacteremia or severe pneumonia requiring active treatment within four weeks prior to the IP administration

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2022-05-08 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
Incidence rate, characteristics, and severity of adverse reactions | up to 52 weeks
  To evaluate the safety of GX-I7 in patients with COVID-19 (rating according to NCI CTCAE v5.0)
Shift from baseline of vital sign | up to 52 weeks
  The number of patients in vital sign shifted from normal or abnormal (NCS) to abnormal (CS)
Shift from baseline of physical examination | up to 52 weeks
  The number of patients in physical examination shifted from normal or abnormal (NCS) to abnormal (CS)
Shift from baseline of hematology | up to 52 weeks
  The number of patients in hematology shifted from normal or abnormal (NCS) to abnormal (CS)
Shift from baseline of blood chemistry | up to 52 weeks
  The number of patients in blood chemistry shifted from normal or abnormal (NCS) to abnormal (CS)
Dose limiting toxicity (DLT) | up to 52 weeks
  The incident rate of DLT

SECONDARY OUTCOMES:
Absolute lymphocyte count (ALC) | up to 3 weeks
  The change of absolute lymphocyte count from baseline
RT-PCR for COVID-19 | up to 52 weeks
  To evaluate the efficacy of GX-I7 in patients with COVID-19
Assessment of clinical improvement by modified early warning score (MEWS) | up to 52 weeks
  Changes of modified early warning score (MEWS) from the baseline after the IP administration [Low-risk (score 0) ~ high-risk (score 3)]
Ordinal scale for clinical improvement (WHO) in each visit | up to 52 weeks
  Changes of ordinal scale for clinical improvement (WHO) from the baseline after the IP administration [Uninfected 0 ~ Dead 8]
The proportion of subjects who have progressed to death or a critical illness | up to 52 weeks
  To evaluate the efficacy of GX-I7 in patients with COVID-19
Immune repertoire | up to 52 weeks
  Changes in the rate of different immune cell types and regulatory T cell in the blood after the IP administration

CONTACTS AND LOCATIONS:
Overall Officials: Minkyu Heo, Study Director — Genexine_Clinical Development Dept.
Locations (1):
- Borame Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No